CLINICAL TRIAL: NCT02497534
Title: Biomarkers in Friedreich's Ataxia
Status: Recruiting | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Children's Miracle Network (Other); National Institutes of Health (NIH) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201500369-N; UL1TR000064 (NIH)
Record Dates: First submitted 2015-07-07; First posted 2015-07-14 (Estimated); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Friedreich's Ataxia
Keywords: ataxia; neuromuscular
MeSH Terms: conditions — Friedreich Ataxia; Ataxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Affected with Friedreich's ataxia: Friedreich's ataxia patients aged 6 to 70 (inclusive). Assessments will include collection of genetic mutation reports, cardiac and exercise MRI, echocardiogram, the Friedreich's Ataxia Rating Scale (FARS), exercise testing with a recombinant bike and/or hand ergometer, pulmonary function testing, and gait analysis. Optional labs include a blood draw, skin biopsy, and/or muscle biopsy.
- Healthy controls: Health controls aged 6 to 70 (inclusive). Assessments will include cardiac and exercise MRI, echocardiogram, the Friedreich's Ataxia Rating Scale (FARS), exercise testing, hand ergometer for exercise testing, pulmonary function testing, gait analysis, and optional blood draws and/or muscle/skin biopsies
- Carriers of Friedreich's ataxia: An obligate carrier aged 18 to 70 (inclusive) of the abnormal Friedreich's ataxia gene by being a parent of a child with Friedreich's ataxia. No assessments are to be conducted. Optional labs include a blood draw, skin biopsy, and/or muscle biopsy.

SUMMARY:
The purpose of this project is to characterize measures of cardiac performance and neuromuscular physiology in FA patients using novel techniques, including echocardiography and magnetic resonance imaging (MRI), metabolic exercise testing, and neurophysiological outcomes.

DETAILED DESCRIPTION:
Friedreich's ataxia (FA) is an autosomal recessive disease caused by a mutation in the frataxin gene (FXN). Although rare, FA is the most common form of hereditary ataxia, affecting 1 in every 50,000 people in the United States. Currently, palliative therapies are the only treatment for FA patients. However, current gene therapy efforts in other neuromuscular diseases have positioned the investigator's research program to extend these discoveries and techniques to FA. As new therapies become available for clinical application, it is crucial to identify non-invasive outcomes measures of cardiac and neuromuscular performance with adequate sensitivity to detect the impact of treatments.

ELIGIBILITY:
Inclusion Criteria:

* Genetic diagnosis of Friedreich's ataxia by DNA sequencing, mutational analysis or protein assay OR be a healthy subject with no evidence of a neuromuscular disorder
* Between the ages of 6 and 70 (inclusive)
* Are able to tolerate metabolic exercise testing
* Are stable on cardiac medication regimen for 3 months prior to screening

Exclusion Criteria:

* Presence of unstable heart disease
* Receipt of cardiac transplant
* Any concurrent medical condition which, in the opinion of the investigators, would make the subject unsuitable for the study

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with Friedreich's ataxia, healthy control subjects, and carriers of Friedreich's ataxia
Sampling Method: Non-Probability Sample
Enrollment: 203 (Estimated)
Dates: Start 2015-09; Primary Completion 2030-06-03 (Estimated); Study Completion 2030-06-03 (Estimated)

PRIMARY OUTCOMES:
Cardiac MRI | Baseline and Follow-Up Visits
  Cardiac MRI will be used to characterize cardiac morphology and function.
Echocardiogram | Baseline and Follow-Up Visits
  Echocardiogram will be used to characterize cardiac morphology and function.
Friedreich's Ataxia Rating Scale (FARS) | Baseline and Follow-Up Visits
  FARS scores describe specific neurological impairments in FA.
Metabolic exercise testing | Baseline and Follow-Up Visits
  Metabolic exercise testing will be performed on either a recumbent bike or hand ergometer and will measure the maximal amount of exercise the subject is able to perform.
Scale for the Assessment and Rating of Ataxia (SARA) | Baseline and Follow-Up Visits
  Clinical scale assessing impairment levels in cerebellar ataxia
Muscle Biopsy | Baseline
  The muscle sample will be used to evaluate Frataxin quantification
Skin Biopsy | Baseline
  Analyses to peripheral tissue used to find out how Friedreich's Ataxia develops.
9-Hole-Peg Test | Baseline and Follow-Up Visits
  Assesses upper extremity function and motor coordination.
Pulmonary Function Testing | Baseline and Follow-Up Visits
  Breathing tests to assess lung strength and function.

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Corti, PT, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States